CLINICAL TRIAL: NCT05316844
Title: The Predictors of Typing Performance in Office Employees With Neck Pain; Neck Disability, Muscle Activity, Posture, and Demographics
Brief Title: Investigation of Predictors of Typing Performance in Office Employees With Neck Pain
Status: Completed | Type: Observational
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Arzu Keskin Aktan, PhD, Asst. Prof., Afyonkarahisar Health Sciences University
Other Study IDs: 2018.282
Record Dates: First submitted 2022-03-29; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Task Performance and Analysis
Keywords: Neck Pain; Office Employees; Task- Specific Performance; Surface Electromyography; Trapezius Muscle; Forward Head Posture; Posture
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Office Employees Group: Office Employees with neck pain
  Interventions: Other: There will be no interventions.

INTERVENTIONS:
Other: There will be no interventions. — Measurements and performance tests were conducted to investigate predictors of work-related performance

SUMMARY:
Determining the predictors that are effective on work performance and preventive approaches to be developed for these predictors must be individual and adaptable to every environment, time, and equipment. In this context, the purpose of the present study was to show the relations between neck disability, Upper Trapezius (UT) muscle activation, posture, and demographic characteristics with typing task performance in office employees who have neck pain by using their equipment in their workplaces.

DETAILED DESCRIPTION:
The present study was conducted to show the relations between neck disability, UT muscle activation, posture, and demographic characteristics with typing task performance in office employees who have neck pain by using their equipment in their workplaces. We hypothesized that UT muscle activation, working posture, and age might be the main predictors of typing performance in office employees with neck pain. For this purpose, full-time office employees who use computers for at least 3 hours a day and have neck pain were invited to the study. Volunteers without any health concern, upper-body injury, and surgery provided informed, written consent to participate in the study.

The participants were given a 10-minute typing task in their working environments, during which right and left UT muscle activation was recorded with Surface Electromyography (sEMG). Work posture was evaluated with Rapid Upper Limb Assessment (RULA) and Forward Head Posture (FHP) was evaluated with Cervical Range of Motion (CROM) Device. Hierarchical Regression Analysis was conducted to examine the predictors of typing performance.

ELIGIBILITY:
Inclusion Criteria:

* Full-time and regular employees in the last 1 year,
* Office employees use computers at desk for at least 3 hours per day
* According to RULA, working in a posture that is above the acceptable level,
* No trauma history
* Non-specific neck pain but no chronic conditions of the cervical spine and upper extremity

Exclusion Criteria:

* Volunteer office employees with neck pain who did not meet the inclusion criteria and those who could not complete the study because of pain, discomfort, etc. were excluded from the study (Dropouts; n=3 because of pain and discomfort, n=1 because of incomplete evaluations not completed on their own will)

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Office workers with neck pain, the sample of the study, were selected from among the people living in Istanbul with the invitation to volunteer.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2022-02-11 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index (NDI) | 10 minutes
  The NDI is a self-reported scale consists of pain intensity, personal care, lifting, reading, headache, concentration, work, driving, sleeping and leisure time activities sections. The total score varies between 0-50 and the increase in total score indicates the increase in the severity of the neck disability: "0-4 no disability, 5-14 mild disability, 15-24 moderate disability, 25-34 severe disability, and ≥35 complete disability".
Maximal Voluntary Isometric Contraction (MVIC) | 10 minutes
  It is measured by Surface Electromyography (sEMG) for upper trapezius muscle. 3 maximum contractions were performed for 6 seconds at the manual muscle testing position. The maximum value among 3 repeats was recorded as Maximal Voluntary Isometric Contraction (MVIC) (mV).
Muscle Activation of Upper Trapezius | 30 minutes
  It is the measurement of the Electromyographic activity of trapezius muscles during typing task. According to The Surface ElectroMyoGraphy for the Non-Invasive Assessment of Muscles Project (SENIAM) recommendations for sensors and sensor placement procedures, sEMG was applied for the upper trapezius muscles while performing the computer task in workplace. The mean values (mV) obtained were normalized according to MVIC. Normalized data (%MVIC) was used in the statistical analysis.
Forward Head Posture | 10 minutes
  The CROM Deluxe is an assessment instrument that lets to measure sagittal, frontal and horizontal plane movements (flexion / extension, lateral flexion, rotation and forward head posture), while resting and also performing a task or work posture.
Rapid Upper Limb Assessment (RULA) | 10 minutes
  The RULA Assessment Tool is used to evaluate the ergonomic risk factors associated with neck, trunk, and upper extremity musculoskeletal disorders (MSD). The RULA considers biomechanical and postural load requirements of job demands. Scores between 1-7 are classified from "acceptable posture" (no action required) to "very high risk" (implement change now).

SECONDARY OUTCOMES:
Body Mass Index (BMI) | 1 minutes
  Body mass index (BMI) is a measurement derived from body mass and body height to evaluate body fat. The BMI is defined as the body mass divided by the square of the body height and is expressed in units of kg/m² (kilogram / square meter). According to the BMI value, it is categorized as underweight (<18.5), normal weight (18.5-24.9), overweight (25-29.9), and Obesity (30 or greater).

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Keskin Aktan, PhD, Principal Investigator — Afyonkarahisar Health Sciences University; Nilufer Keskin Dilbay, MSc, Principal Investigator — Marmara University; Zafer Erden, PhD, Prof, Study Director — Hacettepe University
Locations (1):
- Afyonkarahisar Health Sciences University, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available.